CLINICAL TRIAL: NCT05326074
Title: The Effects of Animal Assisted Therapy in Outpatient Psychiatry Clinics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB Concerns
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00080233
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2022-04

CONDITIONS: Anxiety; Depression; Psychiatric or Mood Diseases or Conditions
Keywords: Animal Assisted Therapy; Loneliness; Depression; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal assisted therapy cohort (Experimental): This arm will be the group that is randomized to receiving animal assisted therapy during outpatient office visits.
  Interventions: Other: Animal assisted therapy cohort
- Control therapy cohort (No Intervention): This arm will be the group that will receive the standard outpatient psychiatric treatment without animal therapy.

INTERVENTIONS:
Other: Animal assisted therapy cohort — A therapy dog will be present in the room during the routine outpatient psychiatric visit.
  Arms: Animal assisted therapy cohort

SUMMARY:
This study will examine whether a session of animal-assisted therapy reduces anxiety levels and improves long-term clinical outcomes of outpatient psychiatric patients in regard to their Generalized Anxiety Disorder (GAD-7), Patient Health Questionnaire (PHQ-9 - Depression assessment), Three Item Loneliness scale (TIL), and Mean Arterial Blood Pressure.

DETAILED DESCRIPTION:
Previous research regarding the value and benefits of Animal-Assisted Therapy (AAT) has often been focused on outcomes within In-Patient settings. One project showed that AATs may offer a decrease in agitated behaviors and an increase in social interactions in people with dementia. Prior research shows a reduction in anxiety when interacting with dogs. These reductions were seen in acutely schizophrenic patients, and General In-patient psychiatric patients. However, prior research has often relied on more obscure assessments that do not offer the validity and reliability seen with the Patient Health Questionnaire (PHQ-9) and the Generalized Anxiety Disorder scale (GAD-7).

Physiological responses have also been measured and show a reduction in blood pressure, norepinephrine, and epinephrine levels within hospitalized patients interacting with AATs. Quality of life and happiness have been shown to improve with the presence of animals. Loneliness has been shown to decrease amongst older adults interacting with AATs once per week. No difference was seen between people interacting with a dog 3 times per week versus once per week, which lends support to the value of a research project where patients may only interact with an AAT once per week.

Other publications regarding AATs focused on the theoretical value and discuss how hypothetically the AATs may be beneficial to patients and their perceived loneliness, stress, anxiety, interactions with others, and depression. These projects offer strong suggestions on future research projects regarding the value of AAT.

The prior research is encouraging to the idea that AATs may be beneficial in out-patient settings to Psychiatrists working with depression and anxiety. Given these prior publications, a desire for further evidence and a project validated by commonly used Psychiatry assessments is proposed here.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient psychiatric patients of Dr. Matt Kern who meet the criteria to be diagnosed with Major Depressive Disorder and/or Generalized Anxiety Disorder via Patient Health Questionnaire (PHQ-9) and/or General Anxiety Disorder (GAD-7)

Exclusion Criteria:

* Prior history of animal related trauma
* Participants that require psychiatric hospitalization during the experiment will have their information excluded from analysis
* Participants who have changes made to any Hypertension / Blood Pressure medications during the experiment will have their Blood Pressure measurements removed from final analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
General Anxiety Disorder-7 (GAD-7) scores | Month 6
  The GAD-7 scores will be collected during the duration of the study and then analyzed upon completion to determine if any significant differences are observed between study arms - a score of 10 or greater on the GAD-7 represents a reasonable cut point for identifying cases of GAD. Cut points of 5, 10, and 15 might be interpreted as representing mild, moderate, and severe levels of anxiety on the GAD-7
Patient Health Questionnaire-9 (PHQ-9) scores | Month 6
  The PHQ-9 scores will be collected during the duration of the study and then analyzed upon completion to determine if any significant differences are observed between study arms - score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression
Three-Item Loneliness Scale (TIL) scores | Month 6
  The TIL scores will be collected during the duration of the study and then analyzed upon completion to determine if any significant differences are observed between study arms - Each question is rated on a 3-point scale: 1 = Hardly Ever; 2 = Some of the Time; 3 = Often. All items are summed to give a total score

SECONDARY OUTCOMES:
Mean Arterial Blood Pressure | Month 6
  Blood Pressure measurements will be taken before and after outpatient visits for all study participants and then compared upon completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Matt Kern, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Animal assisted therapy for heart failure patients — https://doi.org/10.4037/ajcc2007.16.6.575
- See also: Animal-assisted therapy on happiness and life quality of chronic psychiatric patients living in psychiatric residential care homes: a randomized controlled study — https://bmcpsychiatry.biomedcentral.com/articles/10.1186/s12888-020-02980-8

DOCUMENTS (1):
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT05326074/ICF_000.pdf